CLINICAL TRIAL: NCT01194258
Title: A Phase II, Randomized, Double Blind, 2-Way Crossover Safety and Efficacy Study of Subcutaneously Injected Prandial Insulins: Lispro-PH20 or Aspart-PH20 Compared to Insulin Lispro (Humalog®) in Patients With Type 2 Diabetes
Brief Title: Safety/Efficacy Study of Subcutaneously Injected Prandial Insulins Compared to Insulin Lispro Alone in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HALO-117-206
Record Dates: First submitted 2010-08-31; First posted 2010-09-02 (Estimated); Results first posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes Mellitus, Type II
Keywords: Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Lispro; Insulin Aspart; insulin glulisine; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lispro-PH20/Insulin lispro (Experimental): All enrolled participants underwent a titration period of 4 to 6 weeks in which they received 100 units per milliliter (U/mL) insulin glulisine, injected subcutaneously (SC), pre-meals, with doses titrated to each participant individually.
  Next, participants were randomly assigned to 1 of 2 study treatments (Treatment A or B) for the first of two, 3-month treatment cycles. Each participant then received the second treatment for the second cycle.
  Lispro-PH20 (Treatment A): 100 U/mL insulin lispro with 5.0 micrograms per milliliter (µg/mL) recombinant human hyaluronidase PH20 (rHuPH20) (combined: Lispro-PH20), injected SC, pre-meals, with doses titrated to each participant individually.
  Insulin Lispro (Treatment B): 100 U/mL insulin lispro, injected SC, pre-meals, with doses titrated to each participant individually.
  Throughout the study, participants requiring basal insulin used twice daily SC injections of 100 U/mL insulin glargine.
  Interventions: Drug: Insulin lispro; Drug: Recombinant human hyaluronidase PH20; Drug: Insulin glulisine; Drug: Insulin glargine
- Aspart-PH20/Insulin Lispro (Experimental): All enrolled participants underwent a titration period of 4 to 6 weeks in which they received 100 U/mL insulin glulisine, injected SC, pre-meals, with doses titrated to each participant individually.
  Next participants were randomly assigned to 1 of 2 study treatments (Treatment A or B) for the first of two, 3-month treatment cycles. Each participant then received the second treatment for the second cycle.
  Aspart-PH20 (Treatment A): 100 U/mL insulin aspart with 5.0 µg/mL rHuPH20 (combined: Aspart-PH20), injected SC, pre-meals, with doses titrated to each participant individually.
  Insulin lispro (Treatment B): 100 U/mL insulin lispro, injected SC, pre-meals, with doses titrated to each participant individually.
  Throughout the study, participants requiring basal insulin used twice daily SC injections of 100 U/mL insulin glargine.
  Interventions: Drug: Insulin lispro; Drug: Insulin aspart; Drug: Recombinant human hyaluronidase PH20; Drug: Insulin glulisine; Drug: Insulin glargine

INTERVENTIONS:
Drug: Insulin lispro
  Other Names: Lispro; Humalog
Drug: Insulin aspart
  Other Names: Aspart; Novolog
  Arms: Aspart-PH20/Insulin Lispro
Drug: Recombinant human hyaluronidase PH20
  Other Names: rHuPH20; PH20; Hylenex
Drug: Insulin glulisine
  Other Names: Apidra
Drug: Insulin glargine
  Other Names: Lantus

SUMMARY:
The purpose of the study was to compare Humalog (insulin lispro)-recombinant human hyaluronidase PH20 (rHuPH20) or Novolog (insulin aspart)-rHuPH20 to insulin lispro for the treatment of Type 2 diabetes mellitus (T2DM) in basal-bolus therapy.

DETAILED DESCRIPTION:
Criteria for randomization into the study included 1) fasting blood glucose and pre-dinner glucose values in the range of 70 to 140 milligrams per deciliter (mg/dL) approximately 60% of the time for 7 days prior to randomization; 2) 90 minute or 2-hour postprandial blood glucose <220 mg/dL approximately 70% of the time for 7 days prior to randomization; and 3) successfully completing 3 days of 10-point glucose monitoring and have at least 4 self-monitored blood glucose values on all non-10-point monitoring days. Participants that did not meet 1 or more of these criteria during a 4- to 6-week Titration Period were not randomized.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥18 years
* Type 2 diabetes mellitus (T2DM) treated with insulin ≥12 months and prandial insulin (at least 2 meals per day) for ≥2 months
* Body mass index (BMI) of 23.0 to 45.0 kilograms per meter squared (kg/m^2)
* Glycosylated hemoglobin (HbA1C) level 7.0 to 8.5%, inclusive
* Fasting C-peptide <0.6 nanograms per milliliter (ng/mL)
* Willingness to use insulin glargine twice a day as basal insulin for the duration of the study
* Willingness to avoid use of an insulin infusion pump or unblinded continuous glucose monitoring (CGM) during the study

Exclusion Criteria:

* Known or suspected allergy to any component of any of the study drugs
* Exclusive use of pre-mixed insulins
* Use of pramlintide, exenatide, and/or liraglutide within 30 days of screening
* Use of sulfonylureas within two months of screening
* Use of drugs (such as corticosteroids or antimetabolites) that could interfere with the interpretation of study results or are known to cause clinically relevant interference with insulin action, glucose utilization, or recovery from hypoglycemia, during the study or within 30 days of screening
* Recurrent severe hypoglycemia (more than 2 episodes over the last 6 months) or hypoglycemic unawareness, as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Muchmore, M.D., Study Director — Halozyme Therapeutics
Locations (22):
- United States (22):
  - John Muir Physician Network Clinical Research Center, Concord, California
  - Medical Group of Encino, Encino, California
  - AMCR Institute, Inc., Escondido, California
  - Marin Endocrine Care and Research, Greenbrae, California
  - Mills-Peninsula Health Services, San Mateo, California
  - Center for Diabetes and Endocrine Care, Hollywood, Florida
  - Diabetes Research Institute, Miami, Florida
  - Baptist Diabetes Associates, Miami, Florida
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Mid-America Diabetes Associates, Wichita, Kansas
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Medstar Research Institute, Hyattsville, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - International Diabetes Center, Minneapolis, Minnesota
  - Mercury Street Medical, Butte, Montana
  - Desert Endocrinology, Henderson, Nevada
  - Diabetes and Endocrinology Associates, PC, Rudd, North Carolina
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Texas Diabetes and Endocrinology, Round Rock, Texas
  - Cetero Research-San Antonio, San Antonio, Texas
  - West Olympia Internal Medicine, Olympia, Washington
  - University of Washington School of Medicine, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included an open-label titration period of at least 4 weeks and up to 6 weeks prior to randomization at Week 0.
Groups:
- All Enrolled Participants: Prior to randomization, all enrolled participants underwent a titration period of 4 to 6 weeks in which they received 100 U/mL insulin glulisine, injected SC, pre-meals, with doses titrated to each participant individually.
  Participants requiring basal insulin used twice daily SC injections of 100 U/mL insulin glargine.
- Insulin Lispro, Then Lispro-PH20: Participants received a subcutaneous (SC) injection of 100 units per milliliter (U/mL) insulin lispro alone pre-meals for 12 weeks during Treatment Period 1 of the study.
  Then, participants received a SC injection of 100 U insulin lispro and 5 micrograms (µg) recombinant human hyaluronidase PH20 (rHuPH20) (combined: Lispro-PH20) pre-meals for 12 weeks during Treatment Period 2 of the study.
- Lispro-PH20, Then Insulin Lispro: Participants received a SC injection of 100 U/mL insulin lispro and 5 µg rHuPH20 (Lispro-PH20) pre-meals for 12 weeks during Treatment Period 1 of the study.
  Then, participants received a SC injection of 100 U/mL insulin lispro alone pre-meals for 12 weeks during Treatment Period 2 of the study.
- Insulin Lispro, Then Aspart-PH20: Participants received a SC injection of 100 U/mL insulin lispro alone pre-meals for 12 weeks during Treatment Period 1 of the study.
  Then, participants received a SC injection of 100 U/mL insulin aspart and 5 µg rHuPH20 (combined: Aspart-PH20) pre-meals for 12 weeks during Treatment Period 2 of the study.
- Aspart-PH20, Then Insulin Lispro: Participants received SC injection of 100 U/mL insulin aspart and 5 µg rHuPH20 (Aspart-PH20) pre-meals for 12 weeks during Treatment Period 1 of the study.
  Then, participants received a SC injection of 100 U/mL insulin lispro alone pre-meals for 12 weeks during Treatment Period 2 of the study.
Period: Titration Period
Arm/Group | All Enrolled Participants | Insulin Lispro, Then Lispro-PH20 | Lispro-PH20, Then Insulin Lispro | Insulin Lispro, Then Aspart-PH20 | Aspart-PH20, Then Insulin Lispro
Started | 132 | 0 | 0 | 0 | 0
Completed | 121 | 0 | 0 | 0 | 0
Not Completed | 11 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 0
Not completed — Titration failure | 3 | 0 | 0 | 0 | 0
Period: Period 1 (12 Weeks)
Arm/Group | All Enrolled Participants | Insulin Lispro, Then Lispro-PH20 | Lispro-PH20, Then Insulin Lispro | Insulin Lispro, Then Aspart-PH20 | Aspart-PH20, Then Insulin Lispro
Started | 0 (Participants were randomized to the Insulin lispro or an Analog-PH20 group after titration.) | 29 (After the titration phase, 29 participants were randomized to the Insulin lispro/Lispro-PH20 group.) | 30 (After the titration phase, 30 participants were randomized to the Lispro-PH20/Insulin lispro group.) | 29 (After the titration phase, 29 participants were randomized to the Insulin lispro/Aspart-PH20 group.) | 33 (After the titration phase, 33 participants were randomized to the Aspart-PH20/Insulin lispro group.)
Received at Least 1 Dose of Study Drug | 0 | 29 | 30 | 29 | 33
Completed | 0 | 29 | 30 | 29 | 32
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 1
Period: Period 2 (12 Weeks)
Arm/Group | All Enrolled Participants | Insulin Lispro, Then Lispro-PH20 | Lispro-PH20, Then Insulin Lispro | Insulin Lispro, Then Aspart-PH20 | Aspart-PH20, Then Insulin Lispro
Started | 0 | 29 | 30 | 29 | 32
Completed | 0 | 27 | 29 | 29 | 30
Not Completed | 0 | 2 | 1 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants in the study, including those who were enrolled but were not randomized.
Groups:
- All Study Participants: All participants in the study, including those who were enrolled but were not randomized.
Arm/Group | All Study Participants
Number analyzed (Participants) | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (9.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 10
  White | 115
  More than one race | 1
  Unknown or Not Reported | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 113
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 132

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin A1C (HbA1C) at the End of Each Treatment Period
Description: Change in glycosylated hemoglobin A1C (HbA1C) from baseline (Week 0) to end of treatment period (Week 12 and Week 24) is presented. Data are presented by combined treatment group (Lispro-recombinant human hyaluronidase PH20 (PH20) + Aspart-PH20 = Analog-PH20) and combined comparator drug (Insulin lispro from both groups). Least squares (LS) means were calculated from linear contrasts of mixed effects linear models with treatment (Lispro, Aspart), PH20 (yes, no), and treatment sequence as fixed effects and participant within treatment sequence as a random effect.
Time Frame: Baseline, Week 12 and Week 24
Population: All participants who completed both Treatment Period 1 and Treatment Period 2 with evaluable HbA1C data.
Measure: Mean (Standard Deviation); unit: percentage of HbA1C
Groups:
- Analog-PH20: 100 U/mL insulin analog (insulin lispro or insulin aspart) with 5.0 µg/mL rHuPH20, injected SC, pre-meals, with doses titrated to each participant individually, for 12 weeks
- Insulin Lispro: 100 U/mL insulin lispro, injected SC, pre-meals, with doses titrated to each participant individually, for 12 weeks
Arm/Group | Analog-PH20 | Insulin Lispro
Number analyzed (Participants) | 115 | 115
percentage of HbA1C | -0.48 (0.590) | -0.46 (0.571)
Statistical Analysis 1: Comparison: Analog-PH20 vs Insulin Lispro; Approximately 110 participants were planned to be enrolled to allow approximately 88 participants to complete both treatment periods. Assuming a dropout rate of ≤20%, an intra-participant correlation of 0.80, a standard deviation of 1.2, and a true difference of 0, the study would have >90% power to show that either Lispro-PH20 or Aspart-PH20 (each tested separately) was non-inferior to insulin lispro alone with respect to the change from baseline in A1C at the end of each treatment period; Test type: Non-Inferiority or Equivalence — Non-inferiority margin was set at 0.40; p = 0.3876, Mixed Models Analysis; LS Mean difference = -0.04, 95% CI 2-sided [-0.12 to 0.05], Standard Error of Mean 0.041

2. Secondary Outcome: Mean Daily Insulin Dose as Recorded During 10-Point Glucose Monitoring
Description: Mean daily insulin dose as recorded during 10-point glucose monitoring is reported. Blood glucose values were obtained during a total of 3 days during each treatment period (3 days during Week 10 of Treatment Period 1 and 3 days during Week 22 of Treatment Period 2) at the following timepoints: immediately prior to breakfast (fasting), 1 hour (hr) after breakfast, 2 hr after breakfast, immediately prior to lunch, 1 hr after lunch, 2 hr after lunch, immediately prior to dinner, 1 hr after dinner, 2 hr after dinner, and at 03:00. A minimum of 7 determinations were required for each day during the 3 days of 10-point glucose profiles. Prandial insulin doses were also recorded during the 10-point glucose monitoring and the mean daily insulin dose over the 3 days was calculated. Data are presented by combined treatment group (Lispro-PH20 + Aspart-PH20 = Analog-PH20) and combined comparator drug (Insulin Lispro from both cohorts).
Time Frame: Week 10 and Week 22
Population: All participants who completed both Treatment Period 1 and Treatment Period 2 with evaluable insulin dosing data.
Measure: Mean (Standard Deviation); unit: units of Insulin
Arm/Group | Analog-PH20 | Insulin Lispro
Number analyzed (Participants) | 104 | 107
units of Insulin | 122.99 (67.150) | 127.47 (69.483)

3. Secondary Outcome: Percentage of Participants Meeting Glucose Targets at Least 2/3 of the Time
Description: Participants were instructed to monitor their blood glucose levels a minimum of 4 times per day on all non-10-point glucose monitoring days. The number of participants meeting 90-minute postprandial plasma glucose (PPG) targets of <140 and <180 milligrams per deciliter (mg/dL) for at least 2/3 of values was recorded during non-10-point glucose monitoring was recorded. The number of participants was recorded, and the percentage of participants meeting glucose targets was calculated by the number of participants with values meeting the specified target at least 2/3 of the time by the total number of participants analyzed, multiplied by 100. Data is presented by combined treatment group (Lispro-PH20 + Aspart-PH20 = Analog-PH20) and combined comparator drug (Insulin Lispro from both cohorts).
Time Frame: Baseline through Week 24, excluding 10-point glucose monitoring days
Population: Participants in Treatment Period 1 or Treatment Period 2 who received at least 1 dose of study drug and had evaluable postprandial blood glucose data.
Measure: Number; unit: Percentage of participants
Arm/Group | Analog-PH20 | Insulin Lispro
Number analyzed (Participants) | 115 | 115
Percentage of participants
  Overall 90-minute PPG <140 mg/dL | 13.9 | 14.8
  PPG <140 mg/dL for breakfast | 24.3 | 17.4
  PPG <140 mg/dL for lunch | 28.7 | 26.1
  PPG <140 mg/dL for dinner | 13.0 | 15.7
  Overall 90 minute PPG <180 mg/dL | 71.3 | 74.8
  PPG <180 mg/dL for breakfast | 70.4 | 65.2
  PPG <180 mg/dL for lunch | 83.5 | 80.0
  PPG <180 mg/dL for dinner | 67.0 | 70.4

4. Secondary Outcome: Rates of Hypoglycemia at the End of Each Treatment Period
Description: The rate of hypoglycemia, defined as blood glucose levels ≤70 mg/dL and <56 mg/dL, was calculated based on 4 weeks of observation prior to the end of treatment period (that is, Week 12 and Week 24). Data are presented by combined treatment group (Lispro-PH20 + Aspart-PH20 = Analog-PH20) and combined comparator drug (Insulin lispro from both groups). A summary of serious and other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Week 12 and Week 24
Population: All participants who completed both Treatment Period 1 and Treatment Period 2.
Measure: Number; unit: Events per participant per month
Arm/Group | Analog-PH20 | Insulin Lispro
Number analyzed (Participants) | 115 | 115
Events per participant per month
  Blood glucose <70 mg/dL (n=111, n=113) | 7.92 | 7.66
  Blood glucose <56 mg/dL (n=91, n=86) | 1.99 | 1.78

5. Secondary Outcome: Change From Baseline in Body Weight at the End of Each Treatment Period
Description: Change from baseline in body weight at the end of each treatment period (Week 12 and Week 24) is presented. Data are presented by combined treatment group (Lispro-PH20 + Aspart-PH20 = Analog-PH20) and combined comparator drug (Insulin lispro from both cohorts).
Time Frame: Baseline, Week 12 and Week 24
Population: All participants who completed both Period 1 and Period 2 with evaluable body weight data.
Measure: Mean (Standard Deviation); unit: pounds
Groups:
- Insulin-lispro: 100 U/mL insulin lispro, injected SC, pre-meals, with doses titrated to each participant individually, for 12 weeks
Arm/Group | Analog-PH20 | Insulin-lispro
Number analyzed (Participants) | 115 | 115
pounds | 3.35 (5.466) | 3.44 (5.852)

6. Secondary Outcome: Mean Daily PPG Excursions
Description: Participants performed 10-point glucose monitoring for a total of 3 days during each treatment period (3 days during Week 10 of Treatment Period 1 and 3 days during Week 22 of Treatment Period 2). Mean daily PPG excursions during 10-point glucose monitoring for breakfast, lunch, and dinner from Treatment Period 1 or Treatment Period 2 are presented. PPG refers to the change in glucose concentration before to after a meal. Data were collected 1 and 2 hours (hr) after each meal. Data are presented by combined treatment group (Lispro-PH20 + Aspart-PH20 = Analog-PH20) and combined comparator drug (insulin lispro from both cohorts).
Time Frame: Week 10 and Week 22
Population: All participants who completed both Period 1 and Period 2 with evaluable PPG excursion data.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Analog-PH20 | Insulin Lispro
Number analyzed (Participants) | 105 | 107
mg/dL
  1 hr after breakfast excursion (n=105, n=107) | 33.67 (34.480) | 40.38 (30.213)
  2 hr after breakfast excursion (n=105, n=107) | 16.64 (40.463) | 22.94 (33.514)
  1 hr after lunch excursion (n=105, n=106) | 18.47 (35.419) | 27.28 (30.075)
  2 hr after lunch excursion (n=104, n=106) | 20.76 (38.939) | 25.27 (34.288)
  1 hr after dinner excursion (n=104, n=107) | 21.24 (32.807) | 18.09 (28.869)
  2 hr after dinner excursion (n=104, n=107) | 12.72 (35.917) | 15.75 (36.104)

ADVERSE EVENTS:
Groups:
- Titration Period: Prior to randomization, all enrolled participants underwent a titration period of 4 to 6 weeks in which they received 100 units per milliliter (U/mL) insulin glulisine, injected subcutaneously (SC), pre-meals, with doses titrated to each participant individually.
- Insulin Lispro (Lispro-PH20 Cohort): Participants randomized to the Lispro-PH20 cohort.
  Participants received a SC injection of 100 U/mL insulin lispro alone pre-meals for 12 weeks during Treatment Period 1 or 2 of the study.
  Throughout the study, participants requiring basal insulin used twice daily SC injections of 100 U/mL insulin glargine.
- Lispro-PH20: Participants received a SC injection of 100 U/mL insulin lispro with 5 micrograms (μg) rHuPH20 pre-meals for 12 weeks during Treatment Period 1 or 2 of the study.
  Throughout the study, participants requiring basal insulin used twice daily SC injections of 100 U/mL insulin glargine.
- Insulin Lispro (Aspart-PH20 Cohort): Participants randomized to the Aspart-PH20 cohort.
  Participants received a SC injection of 100 U/mL insulin lispro alone pre-meals for 12 weeks during Treatment Period 1 or 2 of the study.
  Throughout the study, participants requiring basal insulin used twice daily SC injections of 100 U/mL insulin glargine.
- Aspart-PH20: Participants received a SC injection of 100 U/mL insulin aspart and 5 μg rHuPH20 pre-meals for 12 weeks during Treatment Period 1 or 2 of the study.
  Throughout the study, participants requiring basal insulin used twice daily SC injections of 100 U/mL insulin glargine.
Arm/Group | Titration Period | Insulin Lispro (Lispro-PH20 Cohort) | Lispro-PH20 | Insulin Lispro (Aspart-PH20 Cohort) | Aspart-PH20
Serious Adverse Events (participants affected / at risk) | 2/132 | 0/59 | 0/59 | 1/60 | 4/62
Other Adverse Events (participants affected / at risk) | 34/132 | 19/59 | 29/59 | 32/60 | 35/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Titration Period (N=132) | Insulin Lispro (Lispro-PH20 Cohort) (N=59) | Lispro-PH20 (N=59) | Insulin Lispro (Aspart-PH20 Cohort) (N=60) | Aspart-PH20 (N=62)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Titration Period (N=132) | Insulin Lispro (Lispro-PH20 Cohort) (N=59) | Lispro-PH20 (N=59) | Insulin Lispro (Aspart-PH20 Cohort) (N=60) | Aspart-PH20 (N=62)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypogonadism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Retinopathy proliferative (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vitreous detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 5 (5) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 3 (3) | 3 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (2) | 2 (2) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Injection site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 3 (4) | 7 (7) | 4 (4)
Influenza (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 4 (4) | 7 (9) | 7 (9) | 3 (3)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Central obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 2 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/53 (0) | 0/10 (0) | 0/10 (0) | 0/14 (0) | 1/15 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 4 (5)
Cluster headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0/79 (0) | 1/38 (1) | 0/38 (0) | 0/34 (0) | 0/34 (0)
Prostatitis (Reproductive system and breast disorders) | 1/79 (1) | 0/38 (0) | 0/38 (0) | 1/34 (1) | 0/34 (0)
Testicular pain (Reproductive system and breast disorders) | 0/79 (0) | 0/38 (0) | 0/38 (0) | 0/34 (0) | 1/34 (1)
Testicular swelling (Reproductive system and breast disorders) | 0/79 (0) | 0/38 (0) | 0/38 (0) | 0/34 (0) | 1/34 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other